CLINICAL TRIAL: NCT06104852
Title: Triage Survey for Neurology Research Eligibility
Acronym: TRIAGE-Neuro
Status: Recruiting | Type: Observational
Sponsor: Adams Clinical (Network)
Responsible Party: Sponsor
Other Study IDs: TRIAGE-Neuro-101
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Participants will be surveyed on demographics, medical history, and current memory and cognitive concerns. Vitals signs, urine drug screen, blood draw may be collected.
Other: Optional Medication Washout — Participants taking memory medications which require a down-taper per the judgment of the study physicians may participate in a medication washout period during study screening.

SUMMARY:
TRIAGE-Neuro is a survey study designed to assess potential participants' eligibility to screen for industry-sponsored neurology clinical trials.

DETAILED DESCRIPTION:
TRIAGE-Neuro is a survey study designed to assess potential participants' eligibility to screen for industry-sponsored neurology clinical trials. Secondary objectives include identifying participant characteristics among the clinical trial-seeking population, identifying the percentage of potential participants currently taking prescribed memory medications that could exclude them from clinical trial participation, examining how changes in prescription memory medications impact performance on cognitive assessments, and identifying the percentage of potential participants whose laboratory results could exclude them from clinical trial participation.

ELIGIBILITY:
Inclusion Criteria:

* Participant and study partner (when applicable) have signed an ICF prior to study-specific procedures being performed.
* Participant and study partner (when applicable) are at least 18 years old.

Exclusion Criteria:

* Participant lacks the language skills or cognitive ability to understand the screening process.
* Participant is pregnant, breast-feeding, or planning to become pregnant.
* History of a clinically significant illness which in the investigator's opinion may impact participant safety or the ability to analyze study results.
* Participant represents an acute suicidal risk, as defined as a "yes" response to ideation on Columbia-Suicide Severity Rating Scale questions 4 or 5, or answer "yes" to behavior questions within 90 days of screening.
* Moderate or severe substance use disorder within 90 days prior to screening, according to DSM-5 criteria that in the investigator's opinion could pose undue risk to the participant.
* Any condition that in the investigator's opinion makes a participant unsuitable for the study.
* Currently employed by Adams Clinical or a first-degree relative of an employee working on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are primarily recruited through social media marketing and referrals from physicians.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of the clinical trial seeking population for whom industry-sponsored clinical research is clinically appropriate, as defined as those who go on to screen for a study. | Up to 52 weeks

SECONDARY OUTCOMES:
Proportion of the clinical trial seeking population who enroll in industry-sponsored studies. | Up to 52 weeks
Change in performance on the Mini Mental Status exam for individuals who discontinue memory medications. | Up to 52 weeks
  Change in performance on the Mini Mental Status exam. This clinician administered cognitive assessment is measured on a scale of 0-30, with higher scores indicating better memory.
Changes in score on the Neuropsychiatric Inventory Questionnaire for individuals who discontinue memory medications. | Up to 52 weeks
  Change in score on the Neuropsychiatric Inventory Questionnaire. This caregiver report includes measures of both severity of neuropsychiatric symptoms (from 0-36) and caregiver distress (0-60). Higher scores indicate greater severity of symptoms and higher levels of caregiver distress.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Copley Clinical, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Berman Clinical, New York, New York